CLINICAL TRIAL: NCT03954522
Title: Evaluation in Children of the Psychological Impact of the Visit of a Hospitalized Relative in ICU
Brief Title: The Visiting Child and His Family in ICU
Acronym: ENVIFAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2018/354
Record Dates: First submitted 2019-04-09; First posted 2019-05-17 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care; Child; Acute Stress Disorder; Post Traumatic Stress Disorder
Keywords: ICU; acute stress; PTSD; child; parent hospitalized
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expérimental (Experimental): psychologist interview and psychometrics scales
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — Child = A clinical interview (recorded, duration approximately 30 min) and a scale of acute stress (IES child) will be performed at 2 times (during the 7 days following the first visit of hospitalized kin and 1 month after the kin was discharged from ICU)
  Accompanying parent/kin = Semi-directive interviews (recorded - duration approximately 30 min) will be performed at the same time as those of the child and will be recorded. The parent/kin will also complete a socio-demographic questionnaire of the family group and a depression anxiety scale (HADS)
  Nursing staff = A semi-directive interview (recorded - duration approximately 30 min) will be performed only once (during the 7 days following the first visit to the hospitalized kin). The caregiver will also complete a socio-demographic questionnaire and a Moral Distress Scale (MDS-R)
  Hospitalized parent = One month after ICU discharge, a depression anxiety scale (HADS) and an acute stress scale (IES) will be performed

SUMMARY:
According to literature, it's difficult to evaluate the impact of the visit of the child in ICU. Currently, no recommendations are available regarding welcome and accompany children who visit their relative hospitalized in ICU. Collaboration between humanities and medical sciences brings to this question a complementary look. Majority of studies investigated the question of the impact of young child ICU visit in a unidirectional linear causality scheme visit = psychopathological impact. The visit of the child in ICU should not be considered as an isolated event whose objective characteristics would be alone vectors of trauma. Contrary, the child visit must be apprehended in relation to the quality of the supports on which the child can count. The investigators hypothesize that children can overcome the visit of a kin hospitalized in ICU if accompanying people can support the child and contain, before and after the visit, the emotions of the child.

ELIGIBILITY:
Inclusion Criteria:

* family groups in which at least one child aged 6 to 14 years having expressed the wish to visit his/her hospitalized relative
* family groups in which the non-hospitalized parent has expressed the wish to accompany his/her child during the visit
* parent hospitalized in ICU is at least 18 years old
* informed consent of children, non-hospitalized and/or hospitalized relatives
* informed consent of the accompanying caregiver

Exclusion Criteria:

* moribund patient
* child unaccompanied by his/her parent/relative during the visit
* non-hospitalized non-French-speaking parent/relative (need to be able to answer the questionnaires)
* child benefiting from a psychological follow-up prior to the hospitalization of his/her parent
* non French-speaking child
* child under 6 years old or older than 14
* hospitalized relative who died before the proposed interview with the child (particular attention will be carry out to the interview conditions. The loss of the hospitalized parent will not allow for an interview on the experience of the visit).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Acute psychotraumatic impact of the visit on the child | 7 days
  Scale of stress (Child IES-R : Impact of Event Scale- Revised) : score calculated on 40 points.
  A score of 17 or greater is considered as clinically relevant
Chronic psychotraumatic impact of the visit on the child | 1 month
  Scale of stress (Child IES-R : Impact of Event Scale- Revised) : score calculated on 40 points.
  A score of 17 or greater is considered as clinically relevant
Psychological experience of the visit for the child | 7 days
  semi directive interview
Parental, family and caregiver support provided to the child during and following the visit | 1 month
  semi directive interviews of caregiver/family
Psychological experience of the visit according the child age | 1 month
  semi directive interview analysed in subgroup: comparison between child aged from 6 to 10 years old versus 11 to 14 years old

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided